CLINICAL TRIAL: NCT01890629
Title: A Multicenter, Randomized, Active-controlled, Parallel Group, Open-label, Exploratory Study to Evaluate the Efficacy on Glucose Variability(MAGE, Glucose SD) and Safety of Initial Combination Therapy of Gemigliptin 50mg q.d., Versus Sitagliptin 100mg q.d., or Glimepiride 2mg q.d. With Metformin 500-1,000mg q.d. in Patients With Type 2 Diabetes
Brief Title: Effects of Gemigliptin Versus Sitagliptin or Glimepiride With Metformin on Glucose Variability(MAGE, Glucose SD) Patients With Type 2 DM(STABLE Study)
Acronym: STABLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL012
Record Dates: First submitted 2013-05-24; First posted 2013-07-02 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — LC15-0444; Metformin; Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gemigliptin + Metformin (Experimental): Gemigliptin 50 mg + Metformin 500 mg to 1000mg for 12 weeks
  Interventions: Drug: Gemigliptin + Metformin / Sitagliptin + Metformin / Glimepiride + Metformin
- Sitagliptin + Metformin (Active Comparator): Sitagliptin 100 mg + Metformin 500 mg to 1000mg for 12 weeks
  Interventions: Drug: Gemigliptin + Metformin / Sitagliptin + Metformin / Glimepiride + Metformin
- Glimepiride + Metformin (Active Comparator): Glimepiride 2 mg + Metformin 500 mg to 1000mg for 12 weeks
  Interventions: Drug: Gemigliptin + Metformin / Sitagliptin + Metformin / Glimepiride + Metformin

INTERVENTIONS:
Drug: Gemigliptin + Metformin / Sitagliptin + Metformin / Glimepiride + Metformin

SUMMARY:
To compare efficacy and safety of initial combination therapy of Gemigliptin versus Sitagliptin or Glimepiride with Metformin on Glucose Variability(MAGE, Glucose SD) in Patients With Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus
* adults aged ≥ 20 and aged ≤ 70 years old
* Patients who had not taken anti diabetes drug for 8 weeks prior to screening visit with HbA1c ≥ 7.5%
* All patients give written informed consent
* Patients applicable to any one of following 3 categories

  1. Patients with surgically induced infertility
  2. Post-menopause woman ≥45 years of age with over 2 years from the last menstruation
  3. Fertile pre-menopause woman or male patients who has consented for use of two or more contraceptive methods at least up to 14 days after final administration of the investigational product to avoid getting pregnant

Exclusion Criteria:

* Patients with Type 1 Diabetes, Patients with Diabetic Ketoacidosis or Diabetic Coma as well as Pre-coma
* Patients with Gestational Diabetes Mellitus or with Secondary Diabetes
* Patients with NYHA Class III, IV Congestive Heart Failure or with Treatment-requiring Arrhythmia
* Patients with Thyroid Dysfunction whose TSH is out of normal range, requiring medication therapy
* Patients with pituitary insufficiency or hypoadrenalism
* Patients whose BMI is less than 20 Kg/m2 or exceeds 40 Kg/m2
* Patients whose Total Bilirubin level is 1.5 times higher than the upper limit of normal range and ALT/AST are > 2.5 times higher than the upper limit of normal range
* Patients currently taking strong CYP3A4 inducers
* Patients currently taking Warfarin, Dicoumar or Digoxin
* Patients currently taking any medication from within 4 weeks before Visit 1 (screening) likely to have significant effects on glycemic control or who require to take such medication
* Patients who had taken anti-obesity drugs within 12 weeks in prior to Visit 1 (screening)
* Subject who had been treated with Insulin or GLP-1 analogue within 6 months before Visit 1 (screening)
* Patients who had participated in other clinical study in the past 3 months before Visit 1 (screening)
* Any other patients whom the investigator considers as inadequate for this study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mean Amplitude Glycemic Excursion | Change of MAGE at Week 12 from baseline

SECONDARY OUTCOMES:
Glucagon | Change of Glucagon at Week 12 from baseline
Active GLP-1 | Change of Active GLP-1 at Week 12 from baseline
CRP | Change of CRP at Week 12 from baseline
Nitrotyrosine | Change of nitrotyrosine at Week 12 from baseline
Glycated albumin | Change of glycated albumin at Week 4 from baseline
Fructosamine | Change of fructosamine at Week 4 from baseline
Glucose Standard Deviation in CGMS data | Change of Glucose SD at Week 12 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: SE Park, Principal Investigator — Kangbuk Samsung Hospital; BW Lee, Principal Investigator — Severance Hospital; JH Jo, Principal Investigator — Seoul St. Mary's Hospital; JH Kim, Principal Investigator — Samsung Medical Center; JH Jung, Principal Investigator — Asan Medical Center
Locations (1):
- Severance hospital, Seoul, South Korea